CLINICAL TRIAL: NCT03949634
Title: Cardiac Safety and Efficacy for Early-stage Breast Cancer Patients Treated With Pegylated Liposomal Doxorubicin（PLD）：an Dynamic Randomized, Positive Control, Open, Multicenter Clinical Study
Brief Title: Cardiac Safety and Efficacy for Early-stage Breast Cancer Patients Treated With Pegylated Liposomal Doxorubicin（PLD)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, chief physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC -DMS- BC-08
Record Dates: First submitted 2019-04-16; First posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 1-dodecylpyridoxal; Docetaxel; Paclitaxel; Doxorubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLD plus CTX sequential docetaxel or PTX (Experimental): pegylated liposomal doxorubicin 35 mg/m2,i.v.,d1, plus cyclophosphamide（CTX） 600 mg/m2,i.v.,d1, sequential docetaxel 100 mg/m2,i.v.,d1, or paclitaxel（PTX） 80mg/m2,i.v.,d1,8,15, once every 21days, for 4 cycles.
  Interventions: Drug: PLD; Drug: CTX; Drug: Docetaxel; Drug: Paclitaxel
- DOX plus CTX sequential docetaxel or PTX (Active Comparator): doxorubicin（DOX） 60 mg/m2,i.v.,d1, plus cyclophosphamide 600 mg/m2,i.v.,d1, sequential docetaxel 100 mg/m2,i.v.,d1, or paclitaxel 80mg/m2,i.v.,d1,8,15, once every 21days, for 4 cycles.
  Interventions: Drug: CTX; Drug: Docetaxel; Drug: Paclitaxel; Drug: Doxorubicin

INTERVENTIONS:
Drug: PLD — pegylated liposomal doxorubicin is 35 mg/m2 intravenously on Days 1 of each 21-day cycle followed by cyclophosphamide.
  Other Names: duomeisu
  Arms: PLD plus CTX sequential docetaxel or PTX
Drug: CTX — cyclophosphamide is 600 mg/m2 intravenously on Days 1 of each 21-day cycle, followed by docetaxel or paclitaxel.
  Other Names: huanlinxianan
Drug: Docetaxel — docetaxel is 100 mg/m2 intravenously on Days 1 of each 21-day cycle.
  Other Names: taisudi
Drug: Paclitaxel — paclitaxel is 80mg/m2 intravenously on Days 1, 8 and 15 of each 21-day cycle.
  Other Names: taisu
Drug: Doxorubicin — doxorubicin is 60 mg/m2 intravenously on Days 1 of each 21-day cycle followed by cyclophosphamide.
  Other Names: ameisu
  Arms: DOX plus CTX sequential docetaxel or PTX

SUMMARY:
This is a randomized, multicenter, open, controlled Post-Marketing Study. 272 early stage female breast cancer patients who were histopathology confirmed with adjuvant chemotherapy indications were enrolled in this study .The subjects will be randomly assigned to one of the two treatment groups at a 1: 1 ratio, and stratified by trastuzumab,age,baseline cardiac risk factors.

DETAILED DESCRIPTION:
Subjects will receive one of two treatment regimens:

Group A: intravenous infusion of pegylated liposomal doxorubicin（PLD） 35 mg/m2, d1; cyclophosphamide 600 mg/m2, intravenous infusion, d1; once every 21days, for 4 cycles. Sequential docetaxel 100 mg/m2, intravenous infusion, d1, or paclitaxel 80mg/m2,intravenous infusion, d1,8,15, once every 21 days, for 4 cycles.

Group B: intravenous infusion of doxorubicin 60 mg/m2, d1; cyclophosphamide 600 mg/m2, intravenous infusion, d1; sequential docetaxel 100 mg/m2, intravenous infusion, d1, or paclitaxel 80mg/m2,intravenous infusion, d1,8,15, once every 21days, for 4 cycles. The primary endpoint is cardiotoxity,the secondary endpoint is 5-year disease-free survival (DFS), 5-year overall survival (OS), and safety: hematology and non hematological toxicity.

ELIGIBILITY:
Inclusion Criteria:

* 1.Subjects had histopathologically confirmed early stage breast cancer with adjuvant chemotherapy treatment evidence;
* 2.Age :18-75years old female;
* 3.High risk of recurrence: axillary lymph node-positive, or axillary lymph node negative with at least one of the following risk factors: triple negative breast cancer, histological grade III, the maximum tumor diameter> 5cm, Ki 67 ≥ 50%, vascular thrombosis positive;
* 4.ECOG score 0-1;
* 5.Expected survival time ≥ 12 months;
* 6.LVEF ≥ 55%;
* 7.Normal ECG, ST segment depression in patients such as coronary angiography, confirm <50% stenosis or incidental premature beats are acceptable;
* 8.Bone Marrow Function: ANC：≥1.5×109/L； PLT：≥100×109/L；Hb: ≥90g/L;
* 9.Liver and renal function:Serum creatinine ≤ normal upper limit (ULN) 1.5times; aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤ULN 2.5times; total bilirubin (TBil) level:≤ ULN 1.5 times, or ≤ ULN 2.5times if Gilbert's syndrome are present;
* 10.Subjects are well-behaved, able to undergo treatment and follow-up, and voluntarily comply with this study and understood the study's research process and signed the informed consent.

Exclusion Criteria:

* 1.New York Heart Association (NYHA) Class II or greater heart failure;
* 2.Severe heart disease or discomfort, including but not limited to: High-risk uncontrolled arrhythmias, atrial tachycardia (heart rate>100/min at rest), significant ventricular arrhythmias (ventricular arrhythmias) or higher, atrioventricular block ([Mobitz 2] or third-degree atrioventricular block); Angina pectoris that needs to be treated with anti-anginal medicine; Valvular heart disease with clinical significance; Electrocardiogram shows transmural myocardial infarction; Uncontrolled high blood pressure(eg: Systolic blood pressure> 180 mmHg or diastolic blood pressure> 100 mmHg);
* 3.Prior received neoadjuvant chemotherapy;
* 4.Severe systemic infection or other serious disease;
* 5.Allergies to chemotherapeutic drugs or their excipients or intolerant patients;
* 6.Other malignant tumors have been found in the past 5 years,except for cured cervical carcinoma in situ, non melanoma of the skin;
* 7.Childbearing age patients who are pregnant or lactation and refusing to take effective contraceptive measures during the trial;
* 8.Received any other test drug treatment or participated in other clinical trials at the same time;
* 9.Other conditions considered to be inappropriate to be enrolled by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
cardiotoxity | 2 years.
  Congestive heart failure with clinical symptoms, or no symptoms but an abnormal LVEF

SECONDARY OUTCOMES:
5-year DFS | 5 years
  5-year disease-free survival rate
5-year OS | 5 years
  5-year overall survival rate
Adverse events (AE) | 5 years
  Incidence and Severity of adverse events according to the CTC AE V4.03

CONTACTS AND LOCATIONS:
Overall Officials: zhimin shao, doctor, Principal Investigator — Fudan University affiliated cancer hospital
Locations (1):
- Fudan University affiliated cancer hospital, Shanghai, China

REFERENCES:
- [Derived] Tang L, He M, Geng C, Fan Z, Ling R, Qiao G, Cai L, Luo T, Jin F, Wang H, Zhang A, Zhang H, Zeng X, Wang X, Jiang M, Wang Z, Shao Z. Pegylated liposomal doxorubicin + cyclophosphamide followed by taxane as adjuvant therapy for early-stage breast cancer: a randomized controlled trial. Oncologist. 2025 Jun 4;30(6):oyaf101. doi: 10.1093/oncolo/oyaf101. PMID 40504550